CLINICAL TRIAL: NCT05209880
Title: An Advance Care Planning Intervention in the Emergency Department: a Randomized Controlled Trial
Brief Title: Advance Care Planning in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Kei Ouchi, Assistant Professor of Emergency Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021P003093
Record Dates: First submitted 2022-01-10; First posted 2022-01-27 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Congestive Heart Failure; Metastatic Cancer; Chronic Kidney Disease Requiring Chronic Dialysis; Chronic Obstructive Pulmonary Disease
Keywords: Advance Care Planning; Palliative Care; Goals of Care; ED GOAL
MeSH Terms: conditions — Heart Failure; Neoplasm Metastasis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The intervention will take place in the emergency department or days after an emergency department visit at home/hospital virtually using zoom or phone by our trained clinicians. At the time of follow-up assessments, participants may also receive additional counseling by our trained clinicians as needed.
  Interventions: Behavioral: ED GOAL
- Control Arm (No Intervention): No intervention will be conducted (standard of care).

INTERVENTIONS:
Behavioral: ED GOAL — The emergency department clinician-led, behavioral intervention (ED GOAL) is designed to engage seriously ill yet clinically stable older adults in the emergency department to address their values and preferences towards end-of-life care with their outpatient clinicians. The intervention consists of an interview to discuss participants' values and preferences for end-of-life care. The participants will receive coaching on how to initiate/re-introduce discussions about end-of-life wishes with their loved ones and outpatient clinicians. The participants' outpatient clinicians will also receive a summary of what participants disclosed via email or mailed letter.
  Arms: Intervention Arm

SUMMARY:
This is a two-armed, parallel-design, pre-/post-intervention assessment study. The investigators will conduct a randomized controlled trial for ED GOAL on a cohort of 120 older adults with serious illness to collect patient-centered outcomes and determine preliminary efficacy on increasing advance care planning engagement (self-reported and/or in the electronic medical record) one month after leaving the emergency department. The investigators will also conduct qualitative interviews with participants of ED GOAL.

DETAILED DESCRIPTION:
ED GOAL, a 6-minute motivational interview conducted in the emergency department (ED), which engages participants to address advance care planning (ACP) conversations with their outpatient clinicians and avoids a time-consuming, sensitive conversation in the time-pressured ED environment. This study is designed to determine the preliminary efficacy of ED GOAL on increasing ACP engagement (by self-report and in the electronic medical record) one month after leaving the ED.

ELIGIBILITY:
Inclusion Criteria:

1. ≥50 years of age AND ≥1 Serious illness* OR ED clinician would not be surprised if patient died in the next 12 months (a validated prognostic sign)
2. English-speaking
3. Capacity to consent

   1. Patient with mild cognitive impairment or mild dementia with capacity to consent (requires a caregiver/study partner to enroll)
   2. Caregiver of patient with moderate/severe dementia with capacity to consent

(*) NYHA Stage III/IV congestive heart failure, chronic obstructive lung disease on home oxygen, chronic kidney disease on dialysis, or metastatic solid tumor cancer. In addition, patients with NYHA Stage I/II congestive heart failure, chronic obstructive lung disease not on home oxygen, chronic kidney disease not on dialysis will be included if recent hospitalization in the last 12 months exists.

Exclusion Criteria:

1. Acute physical or emotional distress
2. Determined by treating or study clinician not to be appropriate
3. Clearly documented goals for medical care** (Unless the treating or study clinician recommends that the intervention is clinically indicated)
4. Delirium (assessed using 3D-CAM)
5. Already enrolled in this study
6. Unable/unwilling to schedule the follow-ups on the calendar
7. Receive both the outpatient care for serious illness and primary care outside of the Mass General Brigham health system

(**)e.g., MOLST, medical order for life-sustaining treatment, documented serious illness conversations in clinician notes within the last 3 months, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kei Ouchi, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shiozawa Y, Morton S, Shirai N, Oelschlager H, Kiernat L, Chary AN, Revette AC, Haimovich A, Desai S, Chang KW, Liu SW, Kennedy M, Schonberg MA, Ouchi K. Exploring Patients' Perceptions of an Advance Care Planning Intervention in the Emergency Department: A Qualitative Study. Acad Emerg Med. 2025 Oct;32(10):1076-1083. doi: 10.1111/acem.70109. Epub 2025 Jul 29. PMID 40729413
- [Derived] Ouchi K, Block SD, Rentz DM, Berry DL, Oelschlager H, Shiozawa Y, Rossmassler S, Berger AL, Hasdianda MA, Wang W, Boyer E, Sudore RL, Tulsky JA, Schonberg MA. Serious Illness Conversations in the Emergency Department for Older Adults With Advanced Illnesses: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jun 2;8(6):e2516582. doi: 10.1001/jamanetworkopen.2025.16582. PMID 40531532
- [Derived] Prachanukool T, Block SD, Berry D, Lee RS, Rossmassler S, Hasdianda MA, Wang W, Sudore R, Schonberg MA, Tulsky JA, Ouchi K. Emergency department-based, nurse-initiated, serious illness conversation intervention for older adults: a protocol for a randomized controlled trial. Trials. 2022 Oct 9;23(1):866. doi: 10.1186/s13063-022-06797-6. PMID 36210436
- See also: National Institutes of Health study record — https://reporter.nih.gov/search/4DqkQh5GPEqNJeo3tJ2fzQ/project-details/10252848

RESULTS

PARTICIPANT FLOW:
Period: 1-Month Follow-up
Arm/Group | Intervention Arm | Control Arm
Started | 70 | 71
Completed | 58 | 56
Not Completed | 12 | 15
Not completed — Spoke with Doctor | 5 | 5
Not completed — Lost to Follow-up | 7 | 9
Not completed — Discontinued | 0 | 1
Period: 3-Month Follow-up
Arm/Group | Intervention Arm | Control Arm
Started | 70 | 71
Completed | 44 | 51
Not Completed | 26 | 20
Not completed — Spoke with Doctor | 17 | 7
Not completed — Lost to Follow-up | 8 | 10
Not completed — Discontinued | 1 | 3
Period: 6-Month Follow-up
Arm/Group | Intervention Arm | Control Arm
Started | 70 | 71
Completed | 35 | 40
Not Completed | 35 | 31
Not completed — Spoke with Doctor | 25 | 14
Not completed — Lost to Follow-up | 9 | 14
Not completed — Discontinued | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 70 | 71 | 141
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean (SD) | 65.6 (8.70) | 67.8 (9.62) | 66.7 (9.21)
Age, Customized [Median (Full Range); unit: years]
  Median [Min, Max] | 66.0 [50.0 to 85.0] | 68.0 [50.0 to 92.0] | 66.0 [50.0 to 92.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 38 | 73
  Male | 35 | 33 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 66 | 70 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 15 | 30
  White | 50 | 53 | 103
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 70 | 71 | 141
Serious Illness [Count of Participants; unit: Participants]
  Solid tumor cancer with metastases or recent hospitalization | 39 | 46 | 85
  COPD on home oxygen or recent hospitalization | 3 | 5 | 8
  CHF (NYHA Class III/IV) or recent hospitalization | 16 | 13 | 29
  CKD on dialysis or recent hospitalization | 10 | 4 | 14
  ED Clinician would not be surprised if patient died in the next 12 months | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Advance Care Planning (ACP) Engagement With Clinicians at One Month
Description: ACP engagement is a one-item question from the validated ACP engagement survey that measures participants' self-reported readiness to discuss their values and preferences with their doctors. The instrument is a 5-point Likert scale ranging from "I have never thought about it (1)" to "I have already done it (5)." A higher score indicates a better outcome.
  Sudore RL, Heyland DK, Barnes DE, Howard M, Fassbender K, Robinson CA, Boscardin J, You JJ. Measuring Advance Care Planning: Optimizing the Advance Care Planning Engagement Survey. J Pain Symptom Manage. 2017 Apr;53(4):669-681.e8. doi: 10.1016/j.jpainsymman.2016.10.367. Epub 2016 Dec 29. PMID: 28042072; PMCID: PMC5730058.
Time Frame: Change from baseline ACP engagement at one month
Population: Some participants did not complete the 1-month follow-up survey. Thus, the number analyzed is different at baseline compared to the 1-month mark.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 70 | 71
score on a scale
  Baseline | 2.84 (1.29) | 2.87 (1.40)
  1-Month: number analyzed (Participants) | 63 | 61
  1-Month | 3.37 (1.07) | 3.32 (1.28)
Statistical Analysis 1: Comparison: Intervention Arm vs Control Arm; Test type: Superiority; p = 0.5835, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Feeling Heard and Understood Survey
Description: A validated instrument for seriously ill patients to report how well they feel heard and understood about their wishes for end-of-life care. This instrument is a 5-point Likert scale: "not at all (1)," "slightly (2)," "moderately (3)," "quite a bit (4)," and "completely (5)." A higher score indicates a better outcome.
  Gramling R, Stanek S, Ladwig S, Gajary-Coots E, Cimino J, Anderson W, Norton SA; AAHPM Research Committee Writing Group, Aslakson RA, Ast K, Elk R, Garner KK, Gramling R, Grudzen C, Kamal AH, Lamba S, LeBlanc TW, Rhodes RL, Roeland E, Schulman-Green D, Unroe KT. Feeling Heard and Understood: A Patient-Reported Quality Measure for the Inpatient Palliative Care Setting. J Pain Symptom Manage. 2016 Feb;51(2):150-4. doi: 10.1016/j.jpainsymman.2015.10.018. Epub 2015 Nov 17. PMID: 26596879.
Time Frame: Baseline & 1, 3, and 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Quality of Communication Survey
Description: A validated instrument to measure the quality of communication about end-of-life care. This instrument is a 10-point Likert scale ranging from "the very worse I could imagine (0)" to "the very best I could imagine (10)". A higher score indicates a better outcome.
  Engelberg RA, Downey L, Curtis JR. Psychometric characteristics of a quality of communication questionnaire assessing communication about end-of-life care. J Palliat Med. 2006 Oct;9(5):1086-98.
Time Frame: Baseline & at 1, 3, and 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Healthcare Utilization
Description: Electronic medical records will be reviewed to find the number of urgent care visits, ED visits, hospitalizations, hospice visits, and outpatient visits.
Time Frame: At 6 and 12 months before and 1, 6, 12 months after enrollment
Reporting Status: Not Posted

5. Secondary Outcome: Mortality
Description: The electronic medical records will be reviewed to find the patients' vital status.
Time Frame: At 1, 3, and 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Qualitative Benefits and Obstacles of Advance Care Planning (ACP) Conversations After ED GOAL
Description: Semi-structured interviews to assess the benefits of ED GOAL and obstacles participants faced in completing more ACP conversations with their outpatient clinicians and loved ones after ED GOAL.
Time Frame: At 1, 3, and/or 6 months
Reporting Status: Not Posted

7. Secondary Outcome: Electronic Medical Record Documentation of Advance Care Planning (ACP) Conversations
Description: The electronic medical record will be reviewed to find clinician documentation of ACP conversations.
Time Frame: At 1, 3, and 6 months
Reporting Status: Not Posted

8. Secondary Outcome: Change in Advance Care Planning (ACP) Engagement With Clinicians at Three Months
Description: as for outcome 1
Time Frame: Change from baseline ACP engagement at three months
Reporting Status: Not Posted

9. Secondary Outcome: Change in Advance Care Planning (ACP) Engagement With Clinicians at Six Months
Description: as for outcome 1
Time Frame: Change from baseline ACP engagement at six months
Reporting Status: Not Posted

10. Secondary Outcome: Participant-reported Completion of Advance Care Planning (ACP) Conversations
Description: Participants are asked if they had completed ACP conversations with their loved ones and clinicians.
Time Frame: At 1, 3, and 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 month, 3 months, and 6 months.
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 4/70 | 4/71
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/71
Other Adverse Events (participants affected / at risk) | 0/70 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT05209880/Prot_SAP_000.pdf